CLINICAL TRIAL: NCT04235868
Title: Clinical Trial of Mesenchymal Stem Cell-derived Pleiotropic Factor in Treating Non-healing Wounds
Brief Title: Mesenchymal Stem Cell-derived Pleiotropic Factor in Treating Non-healing Wounds
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiaobing Fu, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-01
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Mesenchymal Stem Cell-derived Bioactivator for Treating Chronic Wounds
MeSH Terms: interventions — Fibroblast Growth Factors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator)
  Interventions: Biological: fibroblast growth factor
- experimental group (Experimental)
  Interventions: Biological: Stem cell-derived derived pleiotropic factor

INTERVENTIONS:
Biological: Stem cell-derived derived pleiotropic factor — After debridement, the wounds in experimental group apply stem cell-derived lyophilized powder, and use foam dressing to wrap the wound; apply once every 2-3 days.
  Arms: experimental group
Biological: fibroblast growth factor — After debridement, the wounds in control group apply fibroblast growth factor to the wound surface, and use foam dressing to wrap the wound; apply once every 2-3 days.
  Arms: control group

SUMMARY:
Chronic wounds do not heal for prolonged periods of time with the significant financial burden on the healthcare system. It has become increasingly essential to improve our clinical treatments. The most promising potential treatment options rely on stem cell-based therapies. A large body of evidence indicates that mesenchymal stem cells can promote wound closure of chronic wounds in animal models and in preclinical studies. MSCs efficacy depends mostly on their paracrine activity. All the bioactive factors and cytokines in MSCs secretions constitute can be collected in the conditioned medium. In here, stem cell-derived conditioned medium was further made into a lyophilized powder. Patients with chronic wounds were enrolled. The wounds in control group treated with fibroblast growth factor commonly used in clinical practice. The wounds in experimental group treated with lyophilized powder. The effectiveness and safety of lyophilized powder will evaluate for chronic wounds.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of chronic wounds; Male or female over 17; Psychologically stable and able to complete the experimental process. -

Exclusion Criteria:

wound greater than 10cm ×10cm; Exposure to radiation or use of hormones, chemotherapy, growth factor dressings and immunosuppressants within 3 months; Participated in other similar tests within 3 months; Pregnant, or lactating women; Severe infectious disease; Severe heart, liver, and kidney dysfunction; Had a history of cancer -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-20 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
wound healing rate | 1 month
  Original wound area minus unhealed wound area then divided by original wound area

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobing Fu, doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Need to contact the researcher and open sharing after the researcher's consent
Supporting Information: Study Protocol
Time Frame: One year after the experiment
Access Criteria: The way of sharing IPD has not yet been determined